CLINICAL TRIAL: NCT00669162
Title: A Phase I/II Trial of Post-Prostatectomy Radiation Therapy, Hormonal Therapy and Concurrent Docetaxel for High Risk Pathologic T2-T3NO (Tumor-3, Node-0) Prostate Cancer
Brief Title: Postoperative Radiation Therapy, Hormonal Therapy and Concurrent Docetaxel for High Risk Pathologic Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12313
Record Dates: First submitted 2008-04-24; First posted 2008-04-29 (Estimated); Results first posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2018-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Radiotherapy; bicalutamide; Goserelin; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RT, Docetaxel, Hormonal Therapy (Experimental): Radiation Therapy (RT) to 66 Gy in 33 treatment fractions at 2.0 Gy/fx Concurrent Docetaxel (with RT) at 20 mg/m2 weekly x 7 Casodex (50 mg po daily)x 6 months Zoladex (10.8 mg sc q 3 mos x 2) or Lupron (22.5 mg im q 3 mos x 2)
  Interventions: Drug: Docetaxel; Radiation: Radiation Therapy; Drug: Casodex and Zoladex (or Lupron)

INTERVENTIONS:
Drug: Docetaxel — 20mg/m2 IV weekly for 7 weeks
  Other Names: Taxotere
Radiation: Radiation Therapy — 66.0 Gy delivered in 33 daily fractions at 2.0 Gy/fx
Drug: Casodex and Zoladex (or Lupron) — Casodex 50 mg po daily for 6 months, and Zoladex 10.8 mg sc q 3 mos x 2 (or Lupron 22.5 mg im q 3 mos x 2)
  Other Names: Bicalutaminde; Leuprolide

SUMMARY:
Following a radical prostatectomy and lymph node sampling, eligible patients will undergo post-operative radiation therapy, concurrent weekly docetaxel chemotherapy , and hormonal therapy (Casodex daily and Zoladex every 3 months for 2 times or Lupron 22.5 mg im every 3 months for 2 times).

DETAILED DESCRIPTION:
After consent, laboratory and radiologic tests will be done and a baseline questionnaire will be completed. Participants will then be started on the protocol specific hormonal therapy for a total of 6 months. After 2 months of hormone therapy the participants will begin radiation therapy and concurrent docetaxel chemotherapy treatments.

The radiation therapy will be delivered to a total dose of 66.0 Gy at 2.0 Gy/fraction (fx) once daily over 7 weeks, using either a 3-D conformal technique and/or intensity modulated radiation therapy (IMRT).

Participants will receive docetaxel once a week for a total of 7 infusions with concurrent radiation therapy treatments. The weekly dose of docetaxel will be 20 mg/m2. Docetaxel will be given as an intravenous (IV) infusion over 30 minutes within ≤6 hours prior to the radiotherapy treatments.

ELIGIBILITY:
Inclusion Criteria:

* Only those patients with adenocarcinoma of the prostate who have undergone a radical prostatectomy with pelvic lymph node sampling and found to have high risk non-metastatic disease with undetectable, persistent or decreasing post-operative Prostate Specific Antigen (PSA) levels, or who have subsequently experienced a rise in PSA, will be eligible for the trial as described below in the inclusion and exclusion criteria
* Histologically documented adenocarcinoma of the prostate.
* Status post radical prostatectomy with sampling of the pelvic lymph nodes with histologically confirmed adenocarcinoma of the prostate, with the patients falling into either the "adjuvant high risk group" or the "salvage high risk group" as follows:

  * a) "Adjuvant High Risk Group" (undetectable, persistent or decreasing PSA levels before starting therapy) who have NO evidence of metastatic disease (i.e. no clinical symptoms or radiologic evidence) who MUST be able to start RT treatments within 6 months of radical prostatectomy with at least one of the 3 disease features:

    1. Pathologic tumor 2-node 0 (T2N0) disease with positive margins and Gleason score ≥8, or
    2. Pathologic tumor 3a-node 0 T3aN0 disease with extracapsular extension and Gleason Score ≥ 8, or
    3. Pathologic tumor 3b-node 0 T3bN0 disease with any Gleason Score
  * b) "Salvage High Risk Group" are those patients with PSA biochemical failure defined by 2 consecutive increases over baseline PSA levels at least one month apart, who have NO other evidence of metastatic disease (i.e. no clinical symptoms or radiologic evidence), and WITH AT LEAST ONE of the high risk disease features as defined below:

    1. Pathologic T3bN0 disease with any Gleason score, or
    2. Pathologic T2-3aN0 disease with Gleason score ≥ 8,
    3. Pathologic T2-3aN0 disease with PSA doubling time ≤10 months, or
    4. Pathologic T2-3aN0 disease with Pre-radiation therapy PSA level ≥1.0 ng/ml
* Neoadjuvant hormonal therapy prior to radical prostatectomy is allowed, and post-prostatectomy hormonal therapy is allowed as long as it is not within 6 months of protocol treatment
* No prior chemotherapy, or pelvic irradiation
* Karnofsky Performance Status ≥70
* Hematologic parameters must be within the following limits:

  * white blood cell count (WBC) ≥ 3,000
  * Platelet Count ≥ 130,000/ mm3
  * Hemoglobin level ≥ 11.0 g/dl
  * Creatinine ≤ 2.5 g/dl
* Normal liver function defined as the following: Total bilirubin below the upper limit of normal AND AST, ALT, and Alkaline Phosphatase must be within a defined range of eligibility as noted below:

  * Alkaline Phosphatase

    * ≤ ULN - eligible
    * > 1x but ≤1.5x ULN - eligible
    * > 2.5x but ≤ 5x ULN - eligible
    * > 5x ULN - ineligible
  * aspartate aminotransferase (AST) or Alanine Aminotransferase (ALT)

    * ≤ upper limit of normal (ULN) - eligible
    * > 1x but ≤1.5x ULN - eligible
    * > 2.5x but ≤ 5x ULN - ineligible
    * > 5x ULN - ineligible
* Patients with a history of an invasive malignancy within the last 5 years are not eligible for the protocol. Patients with history of benign tumors such as a pituitary macroadenomas, meningiomas, or craniopharyngiomas are eligible as long as the benign tumor is under local control regardless of the time frame. Patients with concurrent adequately treated basal cell or squamous cell carcinoma of the skin are also eligible for the protocol.
* Patients must be informed of the investigative nature of the treatment, must give appropriate informed consent to protocol procedures and must sign an Informed Consent Documentation Form.
* Must not have concomitant medical, psychological or social circumstances which would interfere with compliance with the protocol treatment and follow-up.
* Age ≥ 18 years
* Men of childbearing potential must be willing to consent to using effective contraception while on treatment and for a reasonable period thereafter, which should be for at least 6 months after the completion of protocol therapy

Exclusion Criteria:

* Patients who have received prior chemotherapy, pelvic irradiation or post-prostatectomy androgen ablation within 6 months of protocol therapy.
* Any coexisting medical condition precluding full compliance with the study.
* Patients with active infections or known infection with HIV.
* Psychological, familiar, sociological or geographical conditions which would not permit compliance with the study protocol.
* Known contraindication to dexamethasone (allergic reaction or systemic fungal infection)
* Pre-existing Grade ≥ 1 peripheral neuropathy
* Patients with a history of a hypersensitivity reaction to products containing Polysorbate 80 (Tween 80)

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-08; Primary Completion 2016-08 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xinglei Shen, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RT, Docetaxel, Hormonal Therapy
Started | 27
Completed | 26
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | RT, Docetaxel, Hormonal Therapy
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Can Safely Tolerate and Complete Adjuvant Hormonal Therapy, Radiation Therapy and Docetaxel After a Radical Prostatectomy
Description: Defined as percentage of patients that complete full dose of Radiation Therapy (RT)
Time Frame: 8 Months
Measure: Number; unit: percentage of participants
Arm/Group | RT, Docetaxel, Hormonal Therapy
Number analyzed (Participants) | 27
percentage of participants | 26

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | RT, Docetaxel, Hormonal Therapy
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 3/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RT, Docetaxel, Hormonal Therapy (N=27)
Hypertension (Cardiac disorders) | 1 (1)
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RT, Docetaxel, Hormonal Therapy (N=27)
Rhinitis (Immune system disorders) | 3 (3)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Cardiac disorders) | 2 (2)
Fatigue (General disorders) | 24 (26)
Insomnia (Psychiatric disorders) | 7 (8)
Weight gain (Investigations) | 3 (4)
Weight loss (Investigations) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis radiation (Skin and subcutaneous tissue disorders) | 1 (1)
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Hot flashes (Endocrine disorders) | 19 (21)
Hypothyroidism (Endocrine disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 13 (16)
Dehydration (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 15 (27)
Flatulence (Gastrointestinal disorders) | 1 (1)
Heartburn (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 7 (7)
Proctitis (Gastrointestinal disorders) | 2 (2)
Taste alteration (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2)
Skin infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Edema limbs (General disorders) | 4 (4)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 1 (1)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (6)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bladder pain (Renal and urinary disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Rectal pain (Gastrointestinal disorders) | 2 (2)
Testicular pain (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cystitis (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Urinary frequency (Renal and urinary disorders) | 11 (14)
Urinary incontinence (Renal and urinary disorders) | 3 (3)
Urinary retention (Renal and urinary disorders) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Gynecomastia (Reproductive system and breast disorders) | 1 (1)
Flu-like syndrome (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes